CLINICAL TRIAL: NCT05820477
Title: Improving Self-Regulation and Social Support for Type 1 Diabetes During Emerging Adulthood (FAMS-T1D)
Brief Title: FAMS-T1D Self-Regulation and Social Support for T1D
Acronym: FAMS-T1D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Vanderbilt University Medical Center (Other); University of California, Merced (Other); Children's Hospital Los Angeles (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Cynthia Berg, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 00148660; 1R01DK124719 (NIH)
Record Dates: First submitted 2023-04-07; First posted 2023-04-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
Keywords: emerging adults; social support; goal setting; diabetes distress; HbA1c; self-efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators use mail-in A1c kits for the primary outcome-hemoglobin A1c-and the lab analyzing these samples is masked to participants' assigned condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAMS-T1D (Experimental): Participants will receive FAMS-T1D components (monthly phone coaching and text message support for goals) for 6 months. Support person will receive text messages that are tailored to the goal set by the person with type 1 diabetes.
  All persons with diabetes will receive text messages regarding how to access their HbA1c results and receive links providing information to assist them in self-care behaviors related to their diabetes. All support persons will also receive materials about type 1 diabetes and how to provide helpful support to the person with diabetes.
  Interventions: Behavioral: FAMS-T1D; Behavioral: Digital resources for diabetes
- Digital resources for diabetes (Placebo Comparator): Persons with type 1 diabetes will receive text messages as to how to access their HbA1c results and digital materials related to self-care behaviors for their diabetes. All support persons will receive digital materials about type 1 diabetes and how to provide helpful support to the person with diabetes.
  Interventions: Behavioral: Digital resources for diabetes

INTERVENTIONS:
Behavioral: FAMS-T1D — Behavioral FAMS-T1D FAMS-T1D involves monthly phone coaching that assists individuals in setting specific and time bound diabetes goals with automated text message support to the patient participant and less frequent automated text messages to their support person, if one is enrolled.
  Other Names: Family/friend Activation to Motivate Self-Care for those with Type 1 Diabetes
  Arms: FAMS-T1D
Behavioral: Digital resources for diabetes — Behavioral: Diabetes Resources High quality digital materials about diabetes management will be provided upon enrollment and send to participants quarterly.

SUMMARY:
The goal of this clinical trial is to evaluate how effective the FAMS-T1D intervention is for improving self-regulation (e.g., setting and meeting goals for type 1 diabetes) and social support for meeting those goals for young adults. The main questions that are examined include 1) whether the intervention improves blood glucose, self-management and diabetes distress across time, 2) whether these improvements occur through better self-regulation and social-regulation, 3) whether the intervention improves outcomes for support persons (a friend or family member invited to participate by the person with diabetes) without increasing support burden and 4) whether the intervention improves for persons with diabetes who are on continuous blood glucose monitor their time in range.

DETAILED DESCRIPTION:
This 12-month intervention is an adaptation and expansion of an intervention originally developed for adults with type 2 diabetes (FAMS; NCT02481596) for young adults with type 1 diabetes. FAMS-T1D includes multiple components:

* Monthly coaching sessions (20-30 minutes each) with young adults with type 1 diabetes by phone. The coaching focuses on how to set specific and achievable diabetes goals and to increase helpful and decrease unhelpful family and friend behaviors related to those goals.
* Daily text messages to the person with diabetes to support meeting diabetes goals and engage support that is helpful in meeting those goals.
* Weekly text messages where the person with diabetes responds to how well they have met their goals followed by personalized feedback from the coach.
* The option to invite an adult support person to also receive text messages that assist the support person in providing support that assists the person with diabetes in meeting their goals set in the coaching sessions.

Participants will be randomized to either the intervention or an active control where individuals receive materials relevant to their type 1 diabetes. We plan to enroll 280 persons with diabetes and support persons (optional for persons with diabetes). Persons with type 1 diabetes and their support person (when enrolled) will be randomized together. The study is powered to detect a .5% reduction in hemoglobin A1c. Analyses will examine effects at 6 months (post intervention) and at 12 months (maintenance of effects). The investigators will impute missing data and individuals will be analyzed as randomized irrespective of whether they withdraw or remain in the study following intention-to-treat principals.

ELIGIBILITY:
Inclusion Criteria:

PERSONS WITH DIABETES

* Ages 18-24
* Have a diagnosis of T1D and has been taking insulin for at least one year
* Comfortable sending texts
* Can speak, read, and write in English
* Meets one of the following two criteria: 1) has a most recent A1c value in of 7.5% or higher (prioritizing EHR, next self-report) or missing in EHR) OR 2) screen positive for diabetes distress on the two-item Diabetes Distress Screen (DDS-2).

SUPPORT PERSON

* Can speak, read, and write in either English or Spanish
* Comfortable sending and receiving texts
* Ages 18 and older

Exclusion Criteria:

PERSONS WITH DIABETES:

* Has a condition that would prohibit study completion (intellectual disability, blindness or auditory limitations, severe mental illness)
* Plans to live outside of the country during study period.

SUPPORT PERSON

* Shares a phone with the patient participant.
* Plans to live outside of the country during study period.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c (Person with Diabetes) | Baseline and 6, 9, and 12 months post baseline
  Higher values indicate values more off target. Hemoglobin A1C assessed by mail-in kits from University of Minnesota ARDL
Change in Self-Management (Person with Diabetes) | Baseline and 6, 9, and 12 months post baseline
  Self-care inventory revised, higher values indicate better self-management (values range from 1 to 5)

SECONDARY OUTCOMES:
Diabetes Distress (Person with Diabetes) | Baseline and 6, 9, and 12 months post baseline
  The Diabetes Distress Scale for Adults with Type 1 Diabetes, higher values indicate greater distress (values range from X to X)

OTHER OUTCOMES:
Change in Self-Regulation Failures (Person with Diabetes) | Baseline, and 6, 9, and 12 months post baseline
  Self-regulation failures (outcome and mediator) regarding failures in blood glucose checking ranging from 1 to 5 where higher values indicate greater failures.
Change in Self-Efficacy (Person with Diabetes) | Baseline, and 6, 9, and 12 months post baseline
  Self-efficacy (outcomes and mediator), with scores ranging from 1 to 10 where higher numbers indicate greater self-efficacy.
Change in Goal planning (Person with Diabetes) | Baseline, and 6, 9, and 12 months post baseline
  Goal Planning (outcome and mediator) subscale from the Goal Systems Assessment Battery with scores ranging from 1 to 5 where higher values indicate greater planning.
Change in Disclosure (Person with Diabetes) | Baseline, and 6, 9, and 12 months post baseline
  Disclosure (outcome and mediator) as measured by disclosure subscale with scores ranging from 1 to 5 where higher values indicate greater disclosure to family and friends
Change in Helpful and Harmful Friend and Family Involvement (Person with Diabetes) | Baseline, and 6, 9, and 12 months post baseline
  Change in Helpful (range 1 to 5, higher scores indicate more helpful involvement) and Harmful friend and family involvement (range 1 to 5, higher scores indicate more harmful involvement) (outcome and mediator) as measured by modified FIAD (Mayberry et al., 2019) for type 1 diabetes management.
Change in emotional support (Person with Diabetes) | Baseline, and 6, 9, and 12 months post baseline
  Emotional support (outcome and mediator). Scores range from 1 to 5, higher scores indicate greater emotional support.
Time in range (Person with Diabetes) | Measured continuously from baseline through 12 months post baseline
  Time in range (outcome). For individuals on a continuous blood glucose monitor (CGM) we collect time in range from their monitor. Higher scores indicate greater time spent with blood glucose values in the target range of 70-180 mg/dL.
Change in solicitation of information from patient (support person) | Baseline, and 6, 9, and 12 months post baseline
  Solicitation of information from patient (outcome and mediator), with higher scores reflecting greater solicitation (range 1 to 5).
Change in support burden (support person) | Baseline, and 6, 9, and 12 months post baseline
  Support burden (outcome and mediator), scores range from 0 to 4, higher scores indicate greater burden.
Change in Diabetes Distress (support person) | Baseline, and 6, 9, and 12 months post baseline
  Support Person Diabetes Distress (outcome) with scores ranging from 0 to 4, higher scores indicate greater burden.
Change in Helpful and Harmful Friend and Family Involvement (support person) | Baseline, and 6, 9, and 12 months post baseline.
  Change in helpful (range 1 to 5, higher scores indicate more helpful involvement) and Harmful friend and family involvement (range 1 to 5, higher scores indicate more harmful involvement) (outcome and mediator) as measured by modified FIAD for type 1 diabetes management
Change in emotional support (support person) | Baseline, and 6, 9, and 12 months post baseline
  Emotional support (outcome and mediator). Scores range from 1 to 5, higher scores indicate greater emotional support.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published, de-identified data will be available upon requests made to the principal investigators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study results are posted on clinical trials and outcomes published in a peer-reviewed journal.
Access Criteria: Contact the principal investigator